CLINICAL TRIAL: NCT04639440
Title: Impact of Adipose Tissue in COVID-19 : From Pathophysiology to Therapeutic Perspectives
Brief Title: Impact of Adipose Tissue in COVID-19
Acronym: COVIFAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Other Study IDs: APHP200983; 2020-A02403-36 (Other: ANSM)
Record Dates: First submitted 2020-10-28; First posted 2020-11-20 (Actual); Last update posted 2020-11-20 (Actual); Status verified 2020-10

CONDITIONS: Covid19
Keywords: Adipose tissue; Covid19; SARS-CoV2
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Obese or overweight patients
  Interventions: Other: Adipose tissue
- Patients without overweight
  Interventions: Other: Adipose tissue

INTERVENTIONS:
Other: Adipose tissue — Adipose tissue sampling

SUMMARY:
Overweight or obese patients are particularly exposed to severe forms of COVID-19. Few data suggest that adipose tissue infected with SARS-CoV-2 could be involved in the onset of the cytokine storm seen in severe forms of COVID-19. The aim of this study is to determine the pathogenesis of SARS-CoV-2-infection of adipose tissue. In particular the investigators will study how this virus enters the adipocyte and how it modulates metabolism and inflammation in the adipose tissue. From these data, the investigators hope to determine at the adipose tissue level, original therapeutic targets to modulate the effects of SARS-CoV-2 at the systemic level.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than or equal to 18 years
* All patients who are obese or overweight (> 25 kg/m2) or non-obese (< or = 25 kg/m2) operated for abdominal vascular surgery
* Beneficiary or entitled to a social security scheme (except AME)

Exclusion Criteria:

* Pregnant or breastfeeding woman
* Patient refusal
* Patient deprived of liberty or subject to a legal protection measure (guardianship, curatorship)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Obese and thin patients operated on for abdominal vascular surgery.
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2020-11-23 (Estimated); Primary Completion 2021-11-22 (Estimated); Study Completion 2021-11-23 (Estimated)

PRIMARY OUTCOMES:
Comparison of the expression of ACE2 and TMPRSS2 in the subcutaneous and visceral adipose tissue of obese patients. Determination of cells expressing ACE2 and TMPRSS2 in whole human adipose tissue. | 12 months
  Analysis of the expression of mRNA and ACE2 and TMPRSS2 proteins in the subcutaneous and visceral adipose tissue of normal weight and obese patients

SECONDARY OUTCOMES:
Demonstration of entry and replication of SARS-CoV-2 in human adipose tissue | 12 months
  Infection of human adipocytes in lean and obese subjects by SARS-CoV-2
Consequences of infection with SARS-CoV-2 on the metabolism and inflammatory state of adipose tissue. | 12 months
  Assessment of the expression and secretion of inflammatory cytokines (TNF-α, IL-1 , IL-4 , IL-6 , IL-7 , IL-10 , IL-12 , IL-13 , IL-18 ¸ IL-23, INF-α, INF-β) after infection with SARS-CoV-2 of adipose tissue / adipocytes of thin and obese subjects.
  Evaluation of SARS-CoV-2 infection on the lipolysis of adipose tissue / adipocytes in thin and obese subjects.
Consequences of infection with SARS-CoV-2 on the metabolism and inflammatory state of adipose tissue. | 12 months
  Evaluation of SARS-CoV-2 infection on the lipolysis of adipose tissue / adipocytes in thin and obese subjects.
Effect of SARS-CoV-2 infection of adipose tissue / adipocytes from thin and obese subjects on endoplasmic reticulum (ER) homeostasis. | 12 months
  Study whether infection with SARS-CoV-2 activates the RE stress pathways in adipose tissue
Target endoplasmic reticulum stress to reduce spread of SARS-CoV-2 from adipose tissue | 12 months
  Use of RE stress inhibitors on adipocytes infected with SARS-CoV-2 and assess their effect on the maturation of the virus in infected cells.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier BOURRON, Dr, Principal Investigator — Hôpital Pitié Salpêtrière - Assistance Publique Hôpitaux de Paris
Locations (1):
- Hôpital de la Pitié Salpêtrière, Paris, France